CLINICAL TRIAL: NCT03368378
Title: Impact of Early Dorsal Venous Complex (eDVC) Ligation on Urinary Continence Recovery in Patients Undergoing Robot-assisted Radical Prostatectomy (RARP)
Brief Title: Early DVC Ligation and Urinary Continence Recovery After RARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco Montorsi, MD, FRCS (Hon), Professor and Chairman, Department of Urology Vita e Salute San Raffaele University, Milan, Italy, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eDVCL
Record Dates: First submitted 2017-11-30; First posted 2017-12-11 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radical prostatectomy; deep venous complex ligation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): During robot-assisted radical prostatectomy after the posterior isolation of seminal vesicles, the Retzius space will be accessed and the endopelvic fascia will be incised. The DVC will be identified and incised. The DVC will be then selectively ligated using a V-lok 3/0 barbed suture. After the early DVC isolation, incision and ligation, the bladder neck will be incised and preserved when possible. A posterior nerve sparing approach will be then performed. During apical dissection, the urethral sphincter will be identified and carefully preserved. Posterior reconstruction and anastomosis will be then performed.
  Interventions: Procedure: Early DVC ligation
- Group 2 (Active Comparator): After the posterior isolation of seminal vesicles, the Retzius space will be accessed and the endopelvic fascia will be incised. The bladder neck will be then incised and preserved when possible. An inter-fascial or intra-fascial nerve-sparing technique will be then performed and the posterolateral aspect of the neurovascular bundles will be preserved. The DVC will be then isolated and selectively ligated using a V-lok 3/0 barbed suture. The anterolateral fibers of the neurovascular bundles will be then identified and preserved when possible. During apical dissection, the urethral sphincter will be identified and carefully preserved. Posterior reconstruction and anastomosis will be then performed.
  Interventions: Procedure: Early DVC ligation

INTERVENTIONS:
Procedure: Early DVC ligation — After the posterior isolation of seminal vesicles, the Retzius space will be accessed and the endopelvic fascia will be incised. The DVC will be identified and incised. The DVC will be then selectively ligated using a V-lok 3/0 barbed suture. This approach would allow for the preservation of the external urethral sphincter and for the identification and preservation of the neurovascular bundles that are located in the anterolateral aspect of the prostate. After the early DVC isolation, incision and ligation, the bladder neck will be incised and preserved when possible. A posterior nerve sparing approach will be then performed. During apical dissection, the urethral sphincter will be identified and carefully preserved. Posterior reconstruction and anastomosis will be then performed.

SUMMARY:
The aim of the study is to evaluate the impact of early deep venous complex ligation (eDVCL) in patients affected by clinically localized prostate cancer (PCa) undergoing robot-assisted radical prostatectomy with or without pelvic lymph node dissection. Overall, 312 patients will be randomized to the standard technique vs. eDVCL. The primary endpoint is represented by early urinary continence recovery. The secondary endpoints are perioperative outcomes, erectile function recovery and positive surgical margins.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients, aged between 18 and 80 years old
2. Planned to receive robot-assisted radical prostatectomy for prostate cancer
3. Able to understand and willing to sign a written informed consent document
4. On stable dose of current regular medication for at least 4 weeks prior to trial entry

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

1. Life expectancy of less than 12 months
2. Previous chemotherapy
3. Previous brachytherapy or external beam radiotherapy
4. Preexisting urinary incontinence defined as 1 or more pads per day
5. Unstable cardiovascular disease
6. Congestive Heart Failure (CHF)
7. Clinically significant hepatobiliary or renal disease
8. History of significant CNS injuries within 6 months
9. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Early urinary continence recovery | 4 weeks
  Continence recovery evaluated with the ICIQ-SF questionnaire

SECONDARY OUTCOMES:
Urinary continence recovery | 16 weeks
  Continence recovery evaluated with Continence recovery evaluated with the ICIQ-SF questionnaire
Erectile function recovery | 16 weeks
  Erectile function recovery evaluated with the IIEF questionnaire
Positive surgical margins | 4 weeks
  Positive surgical margins
PSA persistence or biochemical recurrence | 4, 16 and 48 weeks
  Serum PSA levels
Perioperative outcomes | 30 days
  Postoperative complications according to the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided